CLINICAL TRIAL: NCT03815591
Title: Implementation and Dissemination of an Evidence-Based Tobacco Product Use Prevention Videogame Intervention With Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2000023070
Record Dates: First submitted 2019-01-11; First posted 2019-01-24 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Smoking Cessation; Smoking
Keywords: smoking; tobacco; e-cigarettes; flavored tobacco
MeSH Terms: conditions — Smoking Cessation; Smoking; Vaping

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adolescents between ages of 10-16 (Experimental): Adolescents given a pre-post survey to measure the effect of the game and building that into the smokeSCREEN video game to anonymously collect information on players' perspectives, beliefs, attitudes, intentions, social norms, and behaviors around tobacco use, and collaborating with youth programs to pilot test how the game can be implemented in real world settings.
  Interventions: Device: smokeSCREEN web-based game

INTERVENTIONS:
Device: smokeSCREEN web-based game — smokeSCREEN tobacco use reduction/prevention web-based game. The game has 1.5-2 hours of unique game play and focuses on combustible cigarettes, e-cigarettes, and flavored tobacco products. Guided by the social cognitive theory and the theory of planned behavior, smokeSCREEN addresses a range of challenges that teens often face involving peer pressure and the use of tobacco products. Participants are provided access to the smokeSCREEN game through a private, password-protected website link and instructed to complete the game.

SUMMARY:
To examine the effects on participants who play the smokeSCREEN game in that the game will have positive changes in their attitudes, beliefs, knowledge, intentions, behaviors and other outcomes related to smoking and tobacco products.

DETAILED DESCRIPTION:
For this project, the CVS Pharmacy Health Foundation has identified after-school, school, and youth programs nationwide with whom to partner. For this project, the play2PREVENT Lab will provide these programs access to the tobacco use reduction/prevention game that the lab has created (smokeSCREEN). Program and school staff will enroll participants between the ages of 10-16 to play smokeSCREEN during their after school, school, and youth program. Before and after gameplay, participants will answer assessment questions related to their attitudes, beliefs, knowledge, intentions, and behaviors around smoking and tobacco product use. The data will be transmitted electronically via the LimeSurvey data collection platform to the Lab, for further analysis. None of the Lab staff will have contact with participants or after-school/school/youth program coordinators or staff.

ELIGIBILITY:
Inclusion Criteria:

* Anyone with a userID and password.

Exclusion Criteria:

* Does not fit the inclusion criteria

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 560 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in beliefs | baseline
  Participants completed a pre-survey through a secured, data collection website (LimeSurvey Data Collection Software), after they have played the videogame intervention. Fourteen questions were designed from the National Youth Tobacco Survey (2014)13 that focused on beliefs about cigarettes, e-cigarettes, and flavored tobacco were used for the survey. For beliefs, questions had 4-5 choices ranging from strongly disagree to strongly agree or definitely yes to definitely not, or 5 responses ranging from unlikely to very likely.
Changes in beliefs | immediately after game play is completed
  Participants completed a post-survey through a secured, data collection website (LimeSurvey Data Collection Software), after they have played the videogame intervention. Fourteen questions were designed from the National Youth Tobacco Survey (2014)13 that focused on beliefs about cigarettes, e-cigarettes, and flavored tobacco were used for the survey. For beliefs, questions had 4-5 choices ranging from strongly disagree to strongly agree or definitely yes to definitely not, or 5 responses ranging from unlikely to very likely.
Change in knowledge | Baseline
  Participants completed a pre-survey through a secured, data collection website (LimeSurvey Data Collection Software), played the videogame intervention. Fourteen questions were designed from the National Youth Tobacco Survey (2014)13 that focused on knowledge about cigarettes, e-cigarettes, and flavored tobacco were used for the surveys. For knowledge, questions had 3 response choices (yes, not, and not sure).
Change in knowledge | immediately after game play is completed
  Participants completed a post-survey through a secured, data collection website (LimeSurvey Data Collection Software), played the videogame intervention. Fourteen questions were designed from the National Youth Tobacco Survey (2014)13 that focused on knowledge about cigarettes, e-cigarettes, and flavored tobacco were used for the surveys. For knowledge, questions had 3 response choices (yes, not, and not sure).
Change in intentions | Baseline
  Participants will complete a pre-survey through a secured, data collection website (LimeSurvey Data Collection Software), immediately before playing the videogame intervention. Survey questions, adapted from the National Youth and Tobacco Use Survey (FDA, 2018), will assess participants' intention of using cigarettes, e-cigarettes, and flavored tobacco. For questions assessing participants' intention of using tobacco products, response options range from definitely not to definitely yes (4 choices).
Change in behaviors | Immediately after gameplay is completed
  Participants will complete a pre-survey through a secured, data collection website (LimeSurvey Data Collection Software), immediately before playing the videogame intervention. Survey questions, adapted from the National Youth and Tobacco Use Survey (FDA, 2018), will assess participants' intention of using cigarettes, e-cigarettes, and flavored tobacco. For questions assessing participants' intention of using tobacco products, response options range from definitely not to definitely yes (4 choices).
Changes in social norms | Baseline
  Participants will complete a pre-survey through a secured, data collection website (LimeSurvey Data Collection Software), immediately before playing the videogame intervention. Survey questions, adapted from the National Youth and Tobacco Use Survey (FDA, 2018), will assess participants' social norms surrounding the use of cigarettes, ecigarettes, and flavored tobacco. Questions assessing the number of friends/peers who use tobacco products will range from 0 to 4 (including an "I don't know" option). Questions, such as "How would your best friends act toward you if you smoked cigarettes," have response options ranging from very unfriendly to very friendly (4 choices).
Changes in social norms | Immediately after gameplay is completed
  Participants will complete a pre-survey through a secured, data collection website (LimeSurvey Data Collection Software), immediately before playing the videogame intervention. Survey questions, adapted from the National Youth and Tobacco Use Survey (FDA, 2018), will assess participants' social norms surrounding the use of cigarettes, ecigarettes, and flavored tobacco. Questions assessing the number of friends/peers who use tobacco products will range from 0 to 4 (including an "I don't know" option). Questions, such as "How would your best friends act toward you if you smoked cigarettes," have response options ranging from very unfriendly to very friendly (4 choices).

SECONDARY OUTCOMES:
Gameplay satisfaction: post-test survey | immediately after game play is completed
  The post-test survey, administered through a secured, data collection website (LimeSurvey Data Collection Software), will include an additional 10 items on the game intervention experience and satisfaction from items designed for a previous videogame study on sexual risk reduction in young adolescents; 4 response choices ranging from strongly disagree to strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Fiellin, MD, Study Director — Yale University
Locations (1):
- play2PREVENT Lab at the Yale Center for Health & Learning Games, New Haven, Connecticut, United States